CLINICAL TRIAL: NCT01177553
Title: Randomized Clinical Trial: Expectant Management vs. Laser Treatment of Monochorionic Twins With Severe Selective Intrauterine Growth Retardation And Absent or Reverse Diastolic Flow in the Umbilical Artery
Brief Title: Randomized Clinical Trial: Expectant Management vs Laser Treatment of Monochorionic Twins With Severe Selective Intrauterine Growth Retardation and Absent or Reverse Diastolic Flow in the Umbilical Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#105690
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Intrauterine Growth Retardation
Keywords: Intrauterine Growth Retardation in Monochorionic Twins
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery Group (Active Comparator): Patients randomized to surgery will have hospital arrangements (laboratory tests and anesthesia assessment) finalized for a surgery the next day. Patients will sign the informed consent form.
  Patients undergoing surgery will be admitted to Tampa General Hospital and will complete usual hospital admission procedures.
  Interventions: Procedure: selective laser photocoagulation of communicating vessels
- Expectant Management Group (Active Comparator): Patients randomized to expectant management will be referred back to their referring obstetrician of perinatologist and advised to undergo weekly ultrasound examinations including Doppler studies of the umbilical artery and amniotic fluid volume. Fetal growth will be assessed every 2-4 weeks. After 24 weeks patients may undergo frequent ultrasound examinations or fetal heart rate monitoring to assess fetal well being. These ultrasounds will be performed by the patient's perinatologist or obstetrician, and will be reported to the research team on an ongoing basis throughout the pregnancy.
  Interventions: Device: Expected Management

INTERVENTIONS:
Procedure: selective laser photocoagulation of communicating vessels — Antibiotic prophylaxis is initiated within an hour of surgery and continued every 8 hours through the first post-operative day. The use of these medications is safe in pregnancy in the doses and schedules outlined. Surgery will be performed under local anesthesia for the mother using 1% xylocaine with epinephrine at the trocar entry site, and IV sedation. The patient will undergo either SLPCV or UCO depending on her choice. Patients will remain hospitalized for 24-48 hours. All subjects will be monitored during their hospital stay. Any unanticipated adverse events or serious adverse events will be reported to the IRB according to IRB reporting requirements. Prior to discharge from the hospital an investigator will perform a post-procedure ultrasound to assess fetal status
  Other Names: SLPCV
  Arms: Surgery Group
Device: Expected Management — Patients randomized to expectant management will be referred back to their referring obstetrician of perinatologist and advised to undergo weekly ultrasound examinations including Doppler studies of the umbilical artery and amniotic fluid volume. Fetal growth will be assessed every 2-4 weeks. After 24 weeks patients may undergo frequent ultrasound examinations or fetal heart rate monitoring to assess fetal well being. These ultrasounds will be performed by the patient's perinatologist or obstetrician, and will be reported to the research team on an ongoing basis throughout the pregnancy.
  Other Names: expectant management (current accepted treatment)
  Arms: Expectant Management Group

SUMMARY:
Intrauterine growth retardation (IUGR) occurs in approximately 3 to 10% of singleton pregnancies, in 9.1% of all twins and 9.9% of monochorionic twins. IUGR in monochorionic twins typically affects only one of the fetuses (selective IUGR or SIUGR). Spontaneous demise of the SIUGR twin can occur, and may result in concomitant demise (up to 40% risk) or severe neurologic handicap (up to 30% risk) of the other twin. These complications result from exsanguination of the appropriately grown (AGA) twin into the demised SIUGR twin through placental vascular communications.

Because the adverse effects to the AGA twin of the spontaneous demise of the SIUGR twin are mediated through placental vascular anastomoses, we have proposed obliterating such anastomoses via endoscopic fetal surgery. We have developed a technique that allows us to identify the vascular anastomoses present in monochorionic placentas. Briefly, deep AV communications are identified on the surface of the placenta by noting that the terminal end of the artery of one of the fetuses does not have a corresponding returning vein to the same fetus. We have speculated that the separation of the circulations may be of benefit in monochorionic twins affected by SIUGR by preventing the adverse effects that may result from the spontaneous demise of the IUGR twin. Our goal is to evaluate with a randomized clinical trial the outcome of SIUGR managed either expectantly or with SLPCV.

Study procedures will begin with confirmation of the diagnosis and screening criteria at the Qualified Clinical Center. The patient will sign the appropriate consents and then be randomized to her treatment group. Enrollment data will be submitted to the research coordinator in Coordinating Center in Tampa. Expectant management patients will be treated by the referring physicians. Laser patients will be treated at Coordinating Center in Tampa General Hospital or qualified laser center. They may return to the referring center for follow-up. After delivery, outcome data will be sent to the research coordinator in Coordinating Center in Tampa.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 16--24 weeks
* Sonographic evidence of monochorionicity: single placenta, same gender, absent twin-peak sign
* Diagnosis of IUGR present in one twin (fetal weight at or below the 10th percentile for gestational age)
* Persistent absent or reverse-end diastolic flow in the umbilical artery in the SIUGR twin
* Able to provide written informed consent

Exclusion Criteria:

* Patients unwilling to participate in the study, provide consent, or to be followed up
* Presence of twin-twin transfusion syndrome (TTTS) defined as a maximum vertical pocket (MVP) of ≤2 cm in one sac and MVP of ≥8 cm in the other sac.
* Presence of major congenital anomalies (anencephaly, acardia, spina bifida) or intracranial findings in either twin: IVH, porencephalic cysts, ventriculomegaly or other findings suggestive of brain damage.
* Both twins are <10th percentile
* Diastolic flow or intermittently absent end-diastolic flow in the umbilical artery in the SIUGR twin
* Unbalanced chromosomal complement (if known).
* Ruptured or detached membranes
* Placental abruption
* Chorioamnionitis
* Triplets
* Active labor
* Jehovah's witness
* Any other patient deemed inappropriate for the study by the principal investigator
* Placenta previa

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A Quintero, MD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - University of South Florida, Tampa, Florida

REFERENCES:
- [Background] Lin CC, Santolaya-Forgas J. Current concepts of fetal growth restriction: part I. Causes, classification, and pathophysiology. Obstet Gynecol. 1998 Dec;92(6):1044-55. doi: 10.1016/s0029-7844(98)00328-7. PMID 9840574
- [Background] Ananth CV, Vintzileos AM, Shen-Schwarz S, Smulian JC, Lai YL. Standards of birth weight in twin gestations stratified by placental chorionicity. Obstet Gynecol. 1998 Jun;91(6):917-24. doi: 10.1016/s0029-7844(98)00052-0. PMID 9610996
- [Background] Hamilton EF, Platt RW, Morin L, Usher R, Kramer M. How small is too small in a twin pregnancy? Am J Obstet Gynecol. 1998 Sep;179(3 Pt 1):682-5. doi: 10.1016/s0002-9378(98)70064-x. PMID 9757971
- [Background] Dudley DK, D'Alton ME. Single fetal death in twin gestation. Semin Perinatol. 1986 Jan;10(1):65-72. No abstract available. PMID 3764450
- [Background] Fusi L, Gordon H. Twin pregnancy complicated by single intrauterine death. Problems and outcome with conservative management. Br J Obstet Gynaecol. 1990 Jun;97(6):511-6. doi: 10.1111/j.1471-0528.1990.tb02521.x. PMID 2198920
- [Background] Lin IJ, Chen CH, Wang TM, Fu LS, Chi CS. Infants of twin pregnancies with one twin demise in the uterus: a retrospective study. Acta Paediatr Taiwan. 1999 Mar-Apr;40(2):92-6. PMID 10910594
- [Background] Axt R, Hippach M, Mink D, Hendrik HJ, Ertan AK, Schmidt W. Maternal and neonatal outcome in a monochorionic twin pregnancy complicated by single intrauterine demise. Clin Exp Obstet Gynecol. 1999;26(3-4):155-7. PMID 10668142
- [Background] Petersen IR, Nyholm HC. Multiple pregnancies with single intrauterine demise. Description of twenty-eight pregnancies. Acta Obstet Gynecol Scand. 1999 Mar;78(3):202-6. PMID 10078581
- [Background] Burke MS. Single fetal demise in twin gestation. Clin Obstet Gynecol. 1990 Mar;33(1):69-78. PMID 2178843
- [Background] Saito K, Ohtsu Y, Amano K, Nishijima M. Perinatal outcome and management of single fetal death in twin pregnancy: a case series and review. J Perinat Med. 1999;27(6):473-7. doi: 10.1515/JPM.1999.063. PMID 10732306
- [Background] Nicolini U, Poblete A. Single intrauterine death in monochorionic twin pregnancies. Ultrasound Obstet Gynecol. 1999 Nov;14(5):297-301. doi: 10.1046/j.1469-0705.1999.14050297.x. No abstract available. PMID 10623986
- [Background] Kilby MD, Govind A, O'Brien PM. Outcome of twin pregnancies complicated by a single intrauterine death: a comparison with viable twin pregnancies. Obstet Gynecol. 1994 Jul;84(1):107-9. PMID 8008302
- [Background] Adegbite AL, Castille S, Ward S, Bajoria R. Neuromorbidity in preterm twins in relation to chorionicity and discordant birth weight. Am J Obstet Gynecol. 2004 Jan;190(1):156-63. doi: 10.1016/j.ajog.2003.07.004. PMID 14749653
- [Background] Karsdorp VH, van Vugt JM, van Geijn HP, Kostense PJ, Arduini D, Montenegro N, Todros T. Clinical significance of absent or reversed end diastolic velocity waveforms in umbilical artery. Lancet. 1994 Dec 17;344(8938):1664-8. doi: 10.1016/s0140-6736(94)90457-x. PMID 7996959
- [Background] Valcamonico A, Danti L, Frusca T, Soregaroli M, Zucca S, Abrami F, Tiberti A. Absent end-diastolic velocity in umbilical artery: risk of neonatal morbidity and brain damage. Am J Obstet Gynecol. 1994 Mar;170(3):796-801. doi: 10.1016/s0002-9378(94)70285-3. PMID 8141204
- [Background] Gratacos E, Carreras E, Becker J, Lewi L, Enriquez G, Perapoch J, Higueras T, Cabero L, Deprest J. Prevalence of neurological damage in monochorionic twins with selective intrauterine growth restriction and intermittent absent or reversed end-diastolic umbilical artery flow. Ultrasound Obstet Gynecol. 2004 Aug;24(2):159-63. doi: 10.1002/uog.1105. PMID 15287053
- [Background] Huber A, Diehl W, Zikulnig L, Bregenzer T, Hackeloer BJ, Hecher K. Perinatal outcome in monochorionic twin pregnancies complicated by amniotic fluid discordance without severe twin-twin transfusion syndrome. Ultrasound Obstet Gynecol. 2006 Jan;27(1):48-52. doi: 10.1002/uog.2655. PMID 16323150
- [Background] De Lia JE, Cruikshank DP, Keye WR Jr. Fetoscopic neodymium:YAG laser occlusion of placental vessels in severe twin-twin transfusion syndrome. Obstet Gynecol. 1990 Jun;75(6):1046-53. PMID 2342732
- [Background] DeLia JE, Cukierski MA, Lundergan DK, Kochenour NK. Neodymium:yttrium-aluminum-garnet laser occlusion of rhesus placental vasculature via fetoscopy. Am J Obstet Gynecol. 1989 Feb;160(2):485-9. doi: 10.1016/0002-9378(89)90477-8. PMID 2916637
- [Background] DeLia JE, Rogers JG, Dixon JA. Treatment of placental vasculature with a neodymium-yttrium-aluminum-garnet laser via fetoscopy. Am J Obstet Gynecol. 1985 Apr 15;151(8):1126-7. doi: 10.1016/0002-9378(85)90395-3. PMID 4039109
- [Background] Ville Y, Hyett J, Hecher K, Nicolaides K. Preliminary experience with endoscopic laser surgery for severe twin-twin transfusion syndrome. N Engl J Med. 1995 Jan 26;332(4):224-7. doi: 10.1056/NEJM199501263320404. PMID 7808488
- [Background] Quintero RA, Morales WJ, Mendoza G, Allen M, Kalter CS, Giannina G, Angel JL. Selective photocoagulation of placental vessels in twin-twin transfusion syndrome: evolution of a surgical technique. Obstet Gynecol Surv. 1998 Dec;53(12 Suppl):S97-103. doi: 10.1097/00006254-199812010-00001. No abstract available. PMID 9870237
- [Background] Quintero RA, Romero R, Reich H, Goncalves L, Johnson MP, Carreno C, Evans MI. In utero percutaneous umbilical cord ligation in the management of complicated monochorionic multiple gestations. Ultrasound Obstet Gynecol. 1996 Jul;8(1):16-22. doi: 10.1046/j.1469-0705.1996.08010016.x. PMID 8843613
- [Background] Lewi L, Gratacos E, Ortibus E, Van Schoubroeck D, Carreras E, Higueras T, Perapoch J, Deprest J. Pregnancy and infant outcome of 80 consecutive cord coagulations in complicated monochorionic multiple pregnancies. Am J Obstet Gynecol. 2006 Mar;194(3):782-9. doi: 10.1016/j.ajog.2005.09.013. PMID 16522413
- [Background] Robyr R, Yamamoto M, Ville Y. Selective feticide in complicated monochorionic twin pregnancies using ultrasound-guided bipolar cord coagulation. BJOG. 2005 Oct;112(10):1344-8. doi: 10.1111/j.1471-0528.2005.00746.x. PMID 16167936
- [Background] Quintero RA, Bornick PW, Morales WJ, Allen MH. Selective photocoagulation of communicating vessels in the treatment of monochorionic twins with selective growth retardation. Am J Obstet Gynecol. 2001 Sep;185(3):689-96. doi: 10.1067/mob.2001.116724. PMID 11568799
- [Background] Hadlock FP, Harrist RB, Martinez-Poyer J. In utero analysis of fetal growth: a sonographic weight standard. Radiology. 1991 Oct;181(1):129-33. doi: 10.1148/radiology.181.1.1887021.
- [Background] Arduini D, Rizzo G, Mancuso S, Romanini C. Short-term effects of maternal oxygen administration on blood flow velocity waveforms in healthy and growth-retarded fetuses. Am J Obstet Gynecol. 1988 Nov;159(5):1077-80. doi: 10.1016/0002-9378(88)90417-6. PMID 3055996
- [Background] Martinez JM, Bermudez C, Becerra C, Lopez J, Morales WJ, Quintero RA. The role of Doppler studies in predicting individual intrauterine fetal demise after laser therapy for twin-twin transfusion syndrome. Ultrasound Obstet Gynecol. 2003 Sep;22(3):246-51. doi: 10.1002/uog.215. PMID 12942495
- [Background] Quintero RA, Comas C, Bornick PW, Allen MH, Kruger M. Selective versus non-selective laser photocoagulation of placental vessels in twin-to-twin transfusion syndrome. Ultrasound Obstet Gynecol. 2000 Sep;16(3):230-6. doi: 10.1046/j.1469-0705.2000.00265.x. PMID 11169288
- [Background] Quintero R. Diagnostic and Operative Fetoscopy. New York: The Parthenon Publishing Group, 2002.
- [Background] Quintero RA, Dickinson JE, Morales WJ, Bornick PW, Bermudez C, Cincotta R, Chan FY, Allen MH. Stage-based treatment of twin-twin transfusion syndrome. Am J Obstet Gynecol. 2003 May;188(5):1333-40. doi: 10.1067/mob.2003.292. PMID 12748508
- [Background] Saunders NJ, Snijders RJ, Nicolaides KH. Therapeutic amniocentesis in twin-twin transfusion syndrome appearing in the second trimester of pregnancy. Am J Obstet Gynecol. 1992 Mar;166(3):820-4. doi: 10.1016/0002-9378(92)91340-g. PMID 1550147
- [Background] Morales W. Selective photocoagulation of placental vessels in twin-twin transfusion syndrome: outcomes and complications. In: Quintero R, ed. Twin-twin transfusion syndrome. London: Taylor and Francis, Scheduled for publication in 2006.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery Group | Expectant Management Group
Started | 3 | 2
Completed | 2 (data as of March 2009) | 2 (data as of March 2009)
Not Completed | 1 | 0
Not completed — babies not yet 6 months of age | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery Group | Expectant Management Group | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Effects of surgery or expectant management on postnatal neurological morbidity of the AGA baby. The primary comparison will be between SLPCV (selective laser photocoagulation of communicating vessels) and expectant management.
Time Frame: 6 months
Measure: Number; unit: percentage of AGA babies who survived
Arm/Group | Surgery Group | Expectant Management Group
Number analyzed (Participants) | 2 | 2
percentage of AGA babies who survived | 100 | 100

2. Secondary Outcome: Fetal/Neonatal/Infant Survival of the AGA Fetus 6 Months After Birth, Comparing the SLPCV (Selective Laser Photocoagulation of Communicating Vessels) and Expectant Management Groups.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Surgery Group | Expectant Management Group
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No